CLINICAL TRIAL: NCT04069390
Title: evaluatioN de la perfOrMAnce De Capteurs E-textiles
Acronym: NOMADE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: BioSerenity (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2019-A00745-52
Record Dates: First submitted 2019-08-23; First posted 2019-08-28 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-04

CONDITIONS: Healthy Volunteers Without Any Cardiac or Any Neurological Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cardioskin-Neuronaute (Experimental)
  Interventions: Device: CARDIOSKIN - Short record; Device: Cardioskin - long record; Device: Neuronaute - long record; Device: Neuronaute -short record

INTERVENTIONS:
Device: CARDIOSKIN - Short record — A short record (max 2H15) is performed with Cardioskin
Device: Cardioskin - long record — A long record (max 8H) is performed with Cardioskin
Device: Neuronaute - long record — A long record (max 8H) is performed with Neuronaute
Device: Neuronaute -short record — A short record (max 2H15) is performed with Neuronaute

SUMMARY:
The NOMADE study has a dual purpose:

* Test the performance of new types of sensors that are likely to integrate Bioserenity devices and will therefore improve them.
* Test the performance of the sensors of Bioserenity CE devices and their advanced versions

Different EC and non-CE models of Neuronaute and Cardioskin may be tested in this study.

DETAILED DESCRIPTION:
Bioserenity develops innovative solutions, using smart clothing that can be used in hospitals or homes, in short or long term. Without wires, these washable textiles allow, in particular, the measurement of biophysiological signals via a recording box, while allowing the participant the freedom to continue his daily activities.

In order to perfect Bioserenity products, new types of non-invasive sensors will be integrated to offer a new range of multimodal and polygraphic products. Moreover, in order to optimise the already EC devices, they have evolved slightly in terms of textile and software.

Participants will perform at least one recording session with one of the study devices, Neuronaute or Cardioskin. After that, they can hold other meetings if they wish. For this they will not be specially summoned, they will have to volunteer when they wish to participate. The model and type of Bioserenity device (Neuronaute or Cardioskin) may change depending on the session. The recording context may also change. Throughout the duration of the study, whether participants wish to participate regularly or not, they will in all cases be limited to two participation sessions per week. They can stop at any time, without having to justify themselves. The investigation centre will adapt to the availability of the participants and their willingness to participate: the aim is to generate them no constraints.

During recording, subjects may be asked to do small, simple exercises, which differ depending on the recorded signal. Sometimes the exercises can be repeated with a non-invasive device of the market, with minimal risks and constraints, in order to be able to perform a comparison of signals

The principal aim evaluate the performance of Cardioskin or Neuronaute device sensors over short-term recording periods.

The secondary aim is to evaluate the performance of Cardioskin or Neuronaute device sensors over long-term recording periods.

ELIGIBILITY:
Inclusion Criteria:

* Male, female at least 18 years
* Membership of a social security scheme

Exclusion Criteria:

* Minors
* Refusal of consent
* Allergy to one of the components of Bioserenity products, including:Polyamide (other polymers),Polyester,Elasthanne,Polyethylene/polyopropylene (other polymers),Titanium,Silicone,Silver/Copper,Other synthetic materials
* Allergy to one of the components present in commercial electrodes (gel electrode type Kendall 530 or similar; or electrodes type Ag/Agcl; or other electrodes containing in particular: acrylate/polyacrylate, acrylic acid, Impedimed electrodes, etc.)
* Allergy to one of the components in an electroconductive cream for sensors (Elefix, Ten20 and similar biocompatible product)
* Known allergy to one of the components in a commercial EEG helmet (neoprene, elastomer, silicone, etc.)
* Sensory disorders that make the participant insensitive to pain
* Motor or mental disorders that prevent the participant from expressing pain
* Behavioural disorders that make the participant excessively agitated or aggressive
* Person protected

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-07-09 (Actual); Primary Completion 2021-01-09 (Estimated); Study Completion 2021-01-09 (Estimated)

PRIMARY OUTCOMES:
performance sensors evaluation -short record | nearly 2 months after each recruitement session
  signal quality will be assessed as "acceptable" or "not acceptable" for interprétation

SECONDARY OUTCOMES:
performance sensors evaluation -long record | nearly 2 months after each recruitement session
  signal quality will be assessed as "acceptable" or "not acceptable" for interpretation

CONTACTS AND LOCATIONS:
Overall Officials: remy WAHNOUN, Principal Investigator — BioSerenity
Locations (1):
- Institut Du Cerveau Et de La Moelle Epiniere, Paris, France

IPD SHARING:
Plan to Share IPD: No